CLINICAL TRIAL: NCT06314334
Title: A Multicenter, Randomized, Controlled Phase II Screening Study of Combined Sequential Chemotherapy and Radiation Therapies for Early-stage Natural Killer/T-cell Lymphoma (IE/IIE)
Brief Title: Screening Study of Combined Sequential Chemotherapy and Radiation Therapy for Early-stage NK/T-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Rong Tao, Prof., Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHCA-NKT-202301
Record Dates: First submitted 2024-03-08; First posted 2024-03-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Natural Killer/T-Cell Lymphoma, Nasal and Nasal-Type
Keywords: Chemotherapy; Radiation therapy; Immune checkpoint inhibitor; Pegaspargase

STUDY DESIGN:
Intervention Model Description: Participants were stratified according to the NRI prognostic index obtained from the baseline assessment (NRI <2, NRI ≥2) and randomly assigned to three groups receiving different experimental treatments.
  Group A (synchronous treatment group) received 4 cycles of Sintilimab combined with pegaspargase therapy. Concurrently, they received radiotherapy treatment. Group B (sequential treatment group) received 4 cycles of the PGEMOX regimen chemotherapy with sequential radiotherapy.
  Group C (sandwiched radiotherapy group) received 2 cycles of the GELAD regimen chemotherapy initially, followed by radiotherapy and another two cycles GELAD chemotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (synchronous treatment group) (Experimental): Patients received 4 cycles of Sintilimab combined with pegaspargase therapy, with each cycle lasting 3 weeks, for a total of 4 cycles. Concurrently, they received radiotherapy treatment (IMRT, 50-56Gy, starting within 21 days after the first Sintilimab treatment).
  Interventions: Drug: Sintilimab+Pegaspargase; Radiation: IMRT
- Group B (sequential treatment group) (Experimental): Patients received 4 cycles of the PGEMOX regimen chemotherapy. Each cycle lasted 3 weeks, with sequential radiotherapy (IMRT, 50-56Gy) administered within 4 weeks after the last chemotherapy cycle.
  Interventions: Drug: P-GemOx; Radiation: IMRT
- Group C (sandwiched radiotherapy group) (Experimental): Patients received 2 cycles of the GELAD regimen chemotherapy initially, with each cycle lasting 3 weeks. After the second cycle of chemotherapy, radiotherapy (IMRT, 50-56Gy) was administered within 4 weeks. Following the completion of radiotherapy, they received an additional 2 cycles of the GELAD regimen chemotherapy.
  Interventions: Drug: GELAD; Radiation: IMRT

INTERVENTIONS:
Drug: Sintilimab+Pegaspargase — 1. Sintilimab, 200mg intravenous drip, on day 1;
  2. pegaspargase, 2000U/m^2, capped at 3750U, intramuscular, day 1;
  Arms: Group A (synchronous treatment group)
Drug: P-GemOx — 1. pegaspargase 2000U/m^2, capped at 3750U on day 1, intramuscular;
  2. gemcitabine 1.0g/m^2 on day 1 and day 8, intravenous drip;
  3. oxaliplatin 130mg/m^2 on day 1, intravenous drip
  Arms: Group B (sequential treatment group)
Drug: GELAD — 1. gemcitabine 1.0g/m^2 on day 1, intravenous drip;
  2. etoposide 60mg/m^2 on day 1-3, intravenous drip;
  3. pegaspargase 2000U/m^2, capped at 3750U on day 1,intramuscular;
  4. dexamethasone 20mg on day 1-4, intravenous drip.
  Arms: Group C (sandwiched radiotherapy group)
Radiation: IMRT — Intensity modulated radiotherapy (50-56Gy)

SUMMARY:
Extranodal NK/T-cell lymphoma, nasal type (NKTCL) is a common malignant tumor in East Asian populations, often starting in the nasal cavity and spreading to other organs. Associated with EBV infection, NKTCL is aggressive. Early-stage patients typically receive chemo and radiotherapy, with promising outcomes. Recent studies show the potential of immune checkpoint inhibitors in NKTCL treatment. However, optimal treatment sequencing and efficacy remain unclear. This study aims to compare three strategies: (A) Pegaspargase with Sintilimab and radiotherapy; (B) chemo then radiotherapy (PGemOx); (C) sandwich chemoradiotherapy (GELAD). The goal is to identify the best treatment based on 24-month progression-free survival.

DETAILED DESCRIPTION:
Extranodal NK/T-cell lymphoma, nasal type (NKTCL) is a malignant hematological tumor that is common in East Asian populations. The disease typically manifests in the nasal cavity in its early stages and can later involve multiple organs throughout the body. Highly associated with EBV infection, NKTCL is known for its aggressive nature. Currently, early-stage patients usually undergo combined treatment with chemotherapy and radiotherapy. Recent studies have shown that combining chemotherapy and radiotherapy containing asparaginase can achieve a complete remission rate (CR) of over 80%, with long-term survival rates exceeding 70% for patients. In recent years, researchers have found that immune checkpoint inhibitors demonstrate high activity in NKTCL, becoming an important therapeutic option. However, it is worth noting that the optimal sequence of chemotherapy and radiotherapy, as well as the effectiveness of combining radiotherapy with immunotherapy, have not been defined. Studies on different treatment strategies have shown variations in treatment-related adverse reactions and compliance with regimens among patients. However, there is currently no prospective randomized controlled study comparing the efficacy and safety of different strategies. Therefore, it is necessary to identify a treatment strategy with good efficacy and tolerability for patients. This study will stratify early-stage NKTCL patients using the NRI scoring system and randomly assign them to three different treatment strategies: (A) asparaginase combined with Sintilimab and synchronous radiotherapy; (B) sequential chemotherapy (PGemOx) followed by radiotherapy ; (C) chemotherapy (GELAD) with sandwiched chemoradiotherapy, to identify the best or worst treatment strategy based on the 24-month progression-free survival rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the diagnostic criteria for NKTCL (WHO-2016) based on pathological examination.
* Primary lesions located in the upper respiratory and digestive tract such as the nasal cavity, sinuses, nasopharynx, oropharynx, or oral cavity, with clinical staging of IE/IIE based on PET/CT and bone marrow examination according to the Lugano 2014 criteria.
* Evaluated for lymphoma response according to the Lugano 2014 criteria, with at least one measurable lesion or lesion assessable by PET/CT.
* No prior treatment with chemotherapy, radiotherapy, immunotherapy, or biological therapy for lymphoma.
* Age between 18 and 75 years, both genders.
* Eastern Cooperative Oncology Group performance status (ECOG) score of 0-2.
* Must have adequate organ and bone marrow function, defined as follows:

Hematology: Absolute neutrophil count (ANC) ≥1.0×10^9/L, platelet count (PLT) ≥75×10^9/L, hemoglobin (Hb) ≥90g/L; no administration of granulocyte colony-stimulating factor, platelet transfusion, or red blood cell transfusion in the previous 14 days.

Liver function: Total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2×ULN.

Renal function: Serum creatinine (Cr) ≤1.5×ULN. Coagulation function: Plasma fibrinogen ≥1.5g/L. Cardiac function: Left ventricular ejection fraction (LVEF) ≥50%, no acute myocardial infarction, arrhythmia, or atrioventricular conduction block of grade I or above on electrocardiogram.

* Willing to comply with the study protocol, follow-up plan, and laboratory and ancillary investigations.

Exclusion Criteria:

* Patients co-infected with HCV, HIV, or HBV with plasma HBV-DNA >10^3/ml.
* Patients with a history of pancreatitis.
* Patients with acute or systemic infections requiring intravenous antibiotic therapy.
* Patients with severe complications such as hemophagocytic syndrome, DIC, etc.
* Significant organ dysfunction: such as respiratory failure, chronic congestive heart failure with NYHA class ≥2, decompensated liver or renal dysfunction, uncontrolled hypertension and diabetes despite aggressive treatment, and cardiovascular thrombotic or hemorrhagic events in the past 6 months.
* Patients with a history of autoimmune diseases who are not suitable for treatment with immune checkpoint inhibitors.
* Pregnant and lactating women.
* Patients with psychiatric disorders.
* Known allergies to drugs in the chemotherapy regimen.
* Patients with concomitant other tumors requiring surgery or chemotherapy within the past 6 months.
* Currently using other experimental drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS24 | From date of randomization until the date of first documented progression, assessed up to 24 months by the Lugano 2014 response criteria.
  Rate of patients with 24-month progression-free survival

SECONDARY OUTCOMES:
ORR | response rate at 24th week
  Overall response rate
OS | From the time of patient randomization to the end of study, assessed up to 60 months
  Overall survival
EFS | From the time of patient randomization to the end of study, assessed up to 60 months
  Event-free survival
TRAE | From the time of patient randomization to the end of study, assessed up to 60 months
  Treatment-related adverse event related to the study drug or intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rong Tao, MD, Study Chair — Fudan Cancer Hospital
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu Y, Tian S, Xu L, Ma Y, Zhang W, Wang L, Jin L, Liu C, Zhu C, Li Z, Hao S, Zhong H, Ding H, Tao R. GELAD chemotherapy with sandwiched radiotherapy for patients with newly diagnosed stage IE/IIE natural killer/T-cell lymphoma: a prospective multicentre study. Br J Haematol. 2022 Feb;196(4):939-946. doi: 10.1111/bjh.17960. Epub 2021 Nov 21. PMID 34806163
- [Background] Zhang Y, Ma S, Cai J, Yang Y, Jing H, Shuang Y, Peng Z, Li B, Liu P, Xia Z, Xia Y, Gao Y, Chen D, Lin J, Li Q, Xu S, Xu Q, Zhang H, Huang H, Cai Q. Sequential P-GEMOX and radiotherapy for early-stage extranodal natural killer/T-cell lymphoma: A multicenter study. Am J Hematol. 2021 Nov 1;96(11):1481-1490. doi: 10.1002/ajh.26335. Epub 2021 Sep 13. PMID 34449095
- [Background] Wang H, Wang L, Li C, Wuxiao Z, Chen G, Luo W, Lu Y. Pegaspargase Combined with Concurrent Radiotherapy for Early-Stage Extranodal Natural Killer/T-Cell Lymphoma, Nasal Type: A Two-Center Phase II Study. Oncologist. 2020 Nov;25(11):e1725-e1731. doi: 10.1634/theoncologist.2020-0144. Epub 2020 Jul 29. PMID 32627928